CLINICAL TRIAL: NCT01831973
Title: An Open-Label, Single-Arm, Multi-center Phase II Study to Evaluate the Efficacy and Safety of TLC388 in Patients With Advanced/Metastatic Renal Cell Carcinoma
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of TLC388 in Advanced/Metastatic RCC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLC388.3
Record Dates: First submitted 2013-03-27; First posted 2013-04-15 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Advanced/Metastasis Renal Cell Carcinoma
MeSH Terms: interventions — TLC 388

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lipotecan, injection for chemotherapy (Experimental): Patients receive TLC388 (50 mg/m2) given as a 30-minute IV infusion, on Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Lipotecan

INTERVENTIONS:
Drug: Lipotecan
  Other Names: TLC388

SUMMARY:
INVESTIGATIONAL PRODUCT:

TLC388 (Lipotecan*) *Lipotecan is a drug product of TLC388 HCl.

PHASE OF DEVELOPMENT:

Phase II

No. OF PATIENTS:

Approximately 40 (Stage I: 15 evaluable patients, Stage II: 25 evaluable patients)

STUDY OBJECTIVES:

Primary

• To evaluate non-progression disease (non-PD) rate at the end of cycle 6

Secondary

* To evaluate progression free survival (PFS)
* To evaluate overall survival (OS)
* To evaluate the duration of non-PD
* To evaluate objective response rate (ORR; where ORR= CR+PR) and duration
* To evaluate the safety profile of TLC388
* To evaluate change in health-related quality of life (HRQOL) at the end of cycle 6

STUDY DESIGN:

This is a Phase II, open-label, single-arm, multi-centre study to evaluate TLC388 monotherapy in patients with locally advanced and/or metastatic renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
A Phase II, open-label, single-arm, multi-center study to evaluate TLC388 monotherapy in patients with locally advanced and/or metastatic RCC. The study consisted of a Screening/Baseline Period, a Treatment Period and a post-treatment Follow-Up Period for PFS and OS.

Patients were to be recruited at two stages. Stage I recruited 15 evaluable patients, who had completed at least 2 cycles of treatment with one tumor assessment. If ≤ 5 patients did not develop PD at the end of cycle 6 per RECIST, no patients were to be recruited for Stage II and the study was to be closed. If > 5 patients did not develop PD at the end of cycle 6, a total of 40 evaluable patients (additional 25 evaluable patients for Stage II) were to be recruited thereafter.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Adult patients defined by age ≥ 18 years
2. Histologically confirmed Renal cell carcinoma (RCC)
3. Locally advanced or metastatic RCC. Locally advanced RCC: defined as a stage T3/T4 disease, not amenable to curative surgery or radiation therapy, with involvement of renal vein/vena cava/peripelvic and perirenal fat/adrenal gland, or invasion beyond Gerota's fascia. Metastatic RCC: equivalent to Stage IV RCC, according to American Joint Committee on Cancer (AJCC) staging
4. Eastern Collaborative Oncology Group (ECOG) Performance Status of ≤ 2. But for the patient with failure of ≥ 2 prior target therapies, ECOG should be ≤ 1.
5. Documented RCC disease with measurable or non-measurable lesion on imaging by RECIST v1.1 (Response Evaluation Criteria in Solid Tumors) criteria
6. Documented treatment failure of at least 1 prior target therapy (sorafenib, sunitinib pazopanib or other VEGF TKI, bevacizumab, temsirolimus, everolimus or other mTOR inhibitor) for advanced or metastatic RCC. If treatment-naïve, patients with poor prognosis features according to Memorial Sloan-Kettering Cancer Centre (MSKCC) risk criteria are acceptable
7. Any acute or chronic adverse effects of prior therapy have resolved to <Grade 2 as determined by CTCAE v4.0 criteria
8. Laboratory values at screening:

   * Absolute neutrophil count ≥ 1,500 /mm3;
   * Platelets ≥ 100,000 /mm3;
   * Hemoglobin ≥ 9.0 g/dL;
   * Total bilirubin ≤ 1.5 times the upper limit of normal;
   * AST (SGOT) ≤ 2.5 times the upper limit of normal;
   * ALT (SGPT) ≤ 2.5 times the upper limit of normal;
   * Serum creatinine ≤ 2 times the upper limit of normal;

EXCLUSION CRITERIA:

1. Pregnancy or lactation. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrolment. Male and female patients of childbearing potential must agree to use appropriate birth control (barrier methods with spermicides, oral or parenteral contraceptives and/or intrauterine devices) during the entire duration of the study, or the patient must be surgically sterile (with documentation in the patient's medical records)
2. Receipt of any chemotherapy for RCC
3. Had cardiac angioplasty or stenting event, myocardial infarction or unstable angina within 3 months of study entry
4. Persistent QTc >450 ms for males, or >470 ms for females, according to Fridericia's correction
5. Patients with Grade 3 or greater hyponatremia at screening
6. History of Class III or IV congestive heart failure according to New York Heart Association (NYHA) classification
7. History of another malignancy, except for non-basal-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix, and not disease free ≥5 years
8. History or presence of central nervous system (CNS) metastasis or leptomeningeal tumors as documented by CT or MRI scan, analysis of cerebrospinal fluid or neurological exam
9. History of human immunodeficiency virus infection
10. Presence of active, uncontrolled infection
11. Radiotherapy received within 4 weeks prior to baseline
12. Use of any investigational agents within 4 weeks of baseline
13. Major surgery within 4 weeks prior to baseline
14. Receipt of radiotherapy to >25 % of bone marrow
15. Concomitant treatment with, or anticipated use of, pharmaceutical or herbal agents which are potent inhibitors or inducers of cytochrome P450 enzymes (Appendix D1), unless approved by the Sponsor
16. Uncontrolled intercurrent illness that would jeopardize patient safety, or interfere with the objectives of the protocol, or limit patient compliance with study requirements, as determined by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2015-03-19 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Non-progression disease (non-PD) rate at the end of cycle 6 | 6 months
  Non-progression disease rate after cycle 6

SECONDARY OUTCOMES:
Progression free survival (PFS) | 3 years
  Progression free survival
Overall survival (OS) | 3 years
  Overall sruvival
Duration of non-PD | 3 years
  Non-progression disease rate (overall)
Objective response rate (ORR; where ORR= CR+PR) and duration | 3 years
  Objective response rate and duration
Safety profile of TLC388 | 3 years
  Serious/ Adverse Events
Change in health-related quality of life (HRQOL) at the end of cycle 6 | 6 months
  Quality of life after cycle 6

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Yvonne Shi, Study Director — Taiwan Liposome Company
Locations (5):
- Taiwan (5):
  - Chang Gung Memorial Hospital. Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital: LinKou Branch, Taoyuan District